CLINICAL TRIAL: NCT04887987
Title: Effects of Two Exercise Programs (Pilates and Multicomponent) Combined With Photobiomodulation Therapy on Pain Intensity, Postural Balance, Perceived Disability, Kinesiophobia, and Pain-related Fear of Movement in Patients With Chronic Non-specific Low Back Pain (CNLBP): a Randomized, Placebo-controlled Clinical Trial.
Brief Title: Effects of Different Exercise Programs Plus Photobiomodulation on Non-specific Low-back Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Norte do Paraná (Other)
Responsible Party: Principal Investigator, Andreo Fernando Aguiar, Principal investigator, Universidade Norte do Paraná
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Photobiomodulation project
Record Dates: First submitted 2021-05-13; First posted 2021-05-17 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Exercise Training; Photobiomodulation Therapy; Low Back Pain
Keywords: Exercise training; Photobiomodulation therapy; Light-emitting diodes; Low back pain; Perceived disability; kinesiophobia; Pain-related fear of moviment
MeSH Terms: conditions — Low Back Pain; Kinesiophobia | interventions — Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pilates exercise program + active PBMT (PIL+PBMT) (Experimental): Participants will be submitted to a supervised 8-wk mat Pilates exercise program (2 x/week) and will receive active PBMT on the lumbar region (between L1 and L5) 10 min before and after exercise sessions (totaling 20 min), through a device containing 264 LEDs (132 red and 132 infrared.
  Interventions: Other: Pilates training + active PBMT
- Pilates exercise program + sham PBMT (PIL+SHAM) (Sham Comparator): Participants will be submitted to a supervised 8-wk mat Pilates exercise program (2 x/week) and will receive sham PBMT on the lumbar region (between L1 and L5) 10 min before and after exercise sessions (totaling 20 min), through a device containing 264 LEDs (132 red and 132 infrared.
  Interventions: Other: Pilates training + sham PBMT
- Multicomponent exercise program + active PBMT (EX+PBMT) (Experimental): Participants will be submitted to a supervised 8-wk multicomponent exercise program (3 x/week) and will receive active PBMT on the lumbar region (between L1 and L5) imediately before each workout, through a device containing 200 LEDs (100 red and 100 infrared).
  Interventions: Other: Multicomponent training + active PBMT
- Multicomponent exercise program + sham PBMT (EX+SHAM) (Sham Comparator): Participants will be submitted to a supervised 8-wk multicomponent exercise program (3 x/week) and will receive sham PBMT on the lumbar region (between L1 and L5) imediately before each workout, through a device containing 200 LEDs (100 red and 100 infrared).
  Interventions: Other: Multicomponent training + sham PBMT

INTERVENTIONS:
Other: Pilates training + active PBMT — Participants will be submitted to a supervised 8-wk mat Pilates exercise program (2 x/week) and will receive active PBMT on the lumbar region 10 min before and after (totaling 20 min) each workout.
  Arms: Pilates exercise program + active PBMT (PIL+PBMT)
Other: Pilates training + sham PBMT — Participants will be submitted to a supervised 8-wk mat Pilates exercise program (2 x/week) and will receive sham PBMT on the lumbar region 10 min before and after (totaling 20 min) each workout.
  Arms: Pilates exercise program + sham PBMT (PIL+SHAM)
Other: Multicomponent training + active PBMT — Participants will be submitted to a supervised 8-wk multicomponent exercise program (3 x/week) and will receive active PBMT on the lumbar region imediately before each workout.
  Arms: Multicomponent exercise program + active PBMT (EX+PBMT)
Other: Multicomponent training + sham PBMT — Participants will be submitted to a supervised 8-wk multicomponent exercise program (3 x/week) and will receive sham PBMT on the lumbar region imediately before each workout.
  Arms: Multicomponent exercise program + sham PBMT (EX+SHAM)

SUMMARY:
The present project aims to examine the effects of different exercise programs (Pilates and multicomponent) combined with photobiomodulation therapy (PBMT) on pain intensity, postural balance, perceived disability, kinesiophobia, and pain-related fear of movement in patients with chronic non-specific low back pain (CNLBP). It was hypothesized that the exercise programs plus active PBMT would outperform the exercise program alone (sham PBMT) in improving postural balance, and decreasing pain intensity, perceived disability, kinesiophobia, and pain-related fear of movement in patients with CNLBP.

DETAILED DESCRIPTION:
The purpose of this study will be to investigate the effects of two different exercise programs (Pilates and multicomponent) combined with photobiomodulation therapy (PBMT) on pain intensity, postural balance, and psychological aspects in individuals with chronic non-specific low back pain (CNLBP). Participants will be randomized into four groups (n = 20 per group): Pilates exercise program + active PBMT (PIL+PBMT), Pilates exercise program + sham PBMT (PIL+SHAM), multicomponent exercise program + active PBMT (EX+PBMT) and multicomponent exercise program + sham PBMT (EX+SHAM). The PIL+PBMT and PIL+SHAM groups will be submitted to a supervised 8-wk mat Pilates exercise program (2 x/week) and will receive their respective PBMT (active or sham) on the lumbar region (between L1 and L5) 10 min before and after exercise sessions (totaling 20 min), through a device containing 264 LEDs (132 red and 132 infrared. The EX+PBMT and EX+SHAM groups will be submitted to a supervised 8-wk multicomponent exercise program (3 x/week) and will receive their respective PBMT (active or sham) on the lumbar region (between L1 and L5) imediately before each workout, through a device containing 200 LEDs (100 red and 100 infrared). The sham PBMT will be applied with the device turned off. Participants and the two physiotherapists responsible for the assessments and exercise sessions will be blinded to PBMT treatments. The following variables will be assessed at pre and post-training: anthropometric measures, peak pain intensity, postural balance, perceived disability (Oswestry Disability Index [ODI], Roland Morris disability questionnaire [RMDQ]), kinesiophobia (Tampa Scale of kinesiophobia [TSK]), and Pain-related fear of movement (Pain Catastrophizing Scale [PCS]), and Fear Avoidance Beliefs Questionnaire [FABQ]. Statistical analyses were performed using IBM SPSS Statistics for Windows (version 24.0; IBM Corp., Armonk, New York). The baseline characteristics will be analyzed using an unpaired Student's t test. Nonparametric tests will be used due to ordinal data of the dependent variables (pain intensity, ODI, RMDQ, TSK, PCS, and FABQ-Phys). The Wilcoxon signed-rank test will be used to assess within-group changes (from pre-intervention to postintervention), while the Mann-Whitney U test will be used to compare the between-groups changes (relative difference, ∆% = [post - pre]/pre*100) for all dependents variables. The significance level will set at p < 0.05. The effect size (r) for within- and between-groups changes will be considered trivial (0.0-<0.1), small (0.1-<0.3), moderate (0.3-<0.5), and large (≥0.5).

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18-75 years
* Self-report of recurrent (≥ 3 x/week) or continuous episodes of nonspecific low back pain for at least 3 months, comprising the lumbar region between L1-L5

Exclusion Criteria:

* To present a history of musculoskeletal disorders that could affect muscle function
* To make use of medicines that could affect muscle function.
* To present low back pain of specific etiology, such as: tumor, herniated disc, facet syndrome, canal stenosis, among others.
* To have used ergogenic supplements and anabolic steroids for at least six months before study
* To present severe skin diseases in the lumbar region, such as: erysipelas, eczema, dermatitis, psoriasis and urticaria
* To have restrictions for exercises practice considering Physical Activity Readiness Questionnaire (PAR-Q) responses.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Peak pain intensity | Baseline and after 8 weeks
  Pain severity will be determine using a 10-point numerical rating scale (NRS), with extremities designated as 0 (no pain) to 10 (unbearable pain). Participants will be instructed to draw a vertical line at a scale point that best matched their level of pain throughout the day. Pain intensity was recorded at night (between 7 and 8 p.m.) for the first 3 days before the intervention (basal) and the last 3 days after the intervention.
Tampa Scale of kinesiophobia (TSK) | Baseline and after 8 weeks
  The TSK is a 17-item self-report questionnaire designed to assess fear of movement, fear of physical activity, and fear avoidance beliefs in patients with chronic LBP [1, 2]. Each item has a 4-point Likert scale ranging from 0 (strongly disagree) to 4 (strongly agree), with individual scores for items 4, 8, 12, and 16 reversed. The total score is the sum of all items ranging from 17 to 68 points, with higher scores indicating a higher level of kinesiophobia [2].
Fear-Avoidance Beliefs Questionnaire (FABQ-Phys) | Baseline and after 8 weeks
  The FABQ is a patient reported questionnaire which specifically focuses on how a patient's fear avoidance beliefs about physical activity (FABQ-Phys) and work may affect and contribute to their low back pain and resulting disability. The FABQ-Phys has four items with a 6-point Likert scale on each, ranging from 0 (strongly disagree) to 6 (strongly agree) [3, 4]. The total score is the sum of all items ranging from 0 to 24, with a higher score indicating a higher level of fear and avoidance behavior associated with beliefs about how physical activity affects LBP.
Pain Catastrophizing Scale (PCS) | Baseline and after 8 weeks
  PCS is a instrument used for measuring catastrophic thinking related to pain. The PCS is a 13-item scale that measures the effect of LBP on rumination, amplification of pain sensations, and feelings of helplessness to control pain [5]. Each item has a 4-point scale ranging from 0 (not at all) to 4 (all the time), on which the participant indicates their level of thoughts and feelings while they are in pain. The total score is the sum of all items on a scale of 0-52 points, with higher scores indicating a higher level of pain catastrophizing [5].
Oswestry Disability Index (ODI) | Baseline and after 8 weeks
  The ODI is used to assess self-reports of disability caused by LBP [6, 7]. The ODI is made up of 10 sections scored from 0 to 5 points, with the total score ranging from 0 to 50 points [6]. A higher score indicates a higher level of disability [6, 8].
Roland Morris Disability Questionnaire (RMDQ) | Baseline and after 8 weeks
  RMDQ questionnaire is designed to assess self-rated physical disability caused by low back pain. The RMDQ consists of 24 items with scores ranging from 0 to 24 points [6]. A higher score indicates a higher level of disability [6, 8].

SECONDARY OUTCOMES:
Postural balance | Baseline and after 8 weeks
  Postural balance will be assess using a force platform. All participants will performed three attempts at static unipedal standing postures (right and left legs) for 30 s each, with a 1 min rest interval in between. The mean of three attempts will be used for analysis. Participants will be instructed to stand on a platform (barefoot), arms parallel to the trunk, eyes open, and look at a target (circle) on a wall 2.5 m away. Stabilographic analysis of the COP will be used to derive the following balance parameters: area of the COP (A-COP), velocity anteroposterior (Vel AP), and velocity mediolateral (Vel ML).

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Norte do Paraná, Londrina, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hudes K. The Tampa Scale of Kinesiophobia and neck pain, disability and range of motion: a narrative review of the literature. J Can Chiropr Assoc. 2011 Sep;55(3):222-32. PMID 21886284
- [Result] Lundberg M, Styf J, Jansson B. On what patients does the Tampa Scale for Kinesiophobia fit? Physiother Theory Pract. 2009 Oct;25(7):495-506. doi: 10.3109/09593980802662160. PMID 19925172
- [Result] Waddell G, Newton M, Henderson I, Somerville D, Main CJ. A Fear-Avoidance Beliefs Questionnaire (FABQ) and the role of fear-avoidance beliefs in chronic low back pain and disability. Pain. 1993 Feb;52(2):157-168. doi: 10.1016/0304-3959(93)90127-B. PMID 8455963
- [Result] Jacob T, Baras M, Zeev A, Epstein L. Low back pain: reliability of a set of pain measurement tools. Arch Phys Med Rehabil. 2001 Jun;82(6):735-42. doi: 10.1053/apmr.2001.22623. PMID 11387576
- [Result] Roland M, Fairbank J. The Roland-Morris Disability Questionnaire and the Oswestry Disability Questionnaire. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3115-24. doi: 10.1097/00007632-200012150-00006. No abstract available. PMID 11124727